CLINICAL TRIAL: NCT00341588
Title: A Case-Control Study of Testicular Germ Cell Tumors Among U.S. Military Servicemen
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999902113; 02-C-N113
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2020-08-21 (Actual); Status verified 2020-08

CONDITIONS: Testicular Cancer
Keywords: Testicular Cancer; Epidemiology; Testicular Germ Cell Cancer; TGCT; Healthy Volunteer
MeSH Terms: conditions — Testicular Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Cases: Male U.S. serviceman, age 18-45 years old with TGCT
- Controls: Male U.S. serviceman, age 18-45 years old without TGCT

SUMMARY:
The incidence of testicular germ cell tumors (TGCT) has increased during the twentieth century and is of particular concern as it primarily affects young men. It is the most common cancer among U.S. males ages 25-34. The only well-described risk factors are cryptorchism (undescended testis), family history of TGCT, and personal history of TGCT. To better understand the environmental and genetic determinants of TGCT risk, a case-control study will be conducted among members of the U.S. armed forces. The study will include men who have donated a blood sample to the Department of Defense Serum Repository (DoDSR) between 1989 and 2000. All DoDSR donors who have developed GCT will be matched to DoDSR donors who have not developed TGCT. Approximately 1,080 men with TGCT, 1,080 controls, and 2,160 mothers will be included in the study.

The DoDSR serum sample will be tested for organochlorines levels, gonadotropin levels, and viral antibody titres. Each participant will donate a saliva specimen that will be used in an examination of genetic susceptibility. Each participant will also complete a questionnaire concerning a variety of possible risk factors such as physical activity, medical history, medication history, and other risk factors. The mothers of all participants will be invited to participate by completing a questionnaire concerning perinatal exposures and events and by donating a saliva sample.

The three main objectives of this study are to:

* determine whether environmental endocrine modulators (i.e., chlorinated pesticides and polychlorinated biphenyls) are related to risk of GCT and, if so, whether their effects are augmented by other risk factors.
* determine whether genetic susceptibility to GCT exists and to characterize the environmental risk factors related to that susceptibility.
* determine whether there are distinct causes of GCT by relating the tissue structures of the tumors to the risk factors.

DETAILED DESCRIPTION:
The incidence of testicular germ cell tumors (TGCT) has increased during the better part of the twentieth century and is of particular concern as it primarily affects young men. Though the tumor is relatively infrequent in the population as a whole, TGCT is the most common cancer among U.S. males in the age group 15-34 years. Despite the increases in TGCT rates, the etiology is still poorly understood. The only well described risk factors for TGCT are cryptorchism, family history of TGCT and personal history of TGCT. Therefore, in order to understand better the environmental and genetic determinants of TGCT risk, a case-control study will be conducted among members of the U.S. Armed Forces. The study will include men who have donated a blood sample to the Department of Defense Serum Repository (DoDSR) between the years 1989 and 2003. All DoDSR donors who have developed GCT will be matched to DoDSR donors who have not developed TGCT.

A total of 1682 servicemen were enrolled in the study; 754 cases and 928 controls. Of these participants, 1303 men (77%, 590 cases, 713 controls) donated buccal cell samples. In addition to the servicemen, a total of 1090 mothers of servicemen were enrolled and 952 (87%) provided a buccal specimen. The DoDSR serum samples have been assayed for levels of organochlorines pesticides, polychlorinated biphenyl congeners, insulin-like growth factors and gonadotropins and steroid hormones. DNA isolated from the buccal cell specimens have thus far been genotyped for polymorphysms in the hormone metabolism and immune function pathway, immune function pathway, insulin-like growth factor pathway and for single nucleotide polymorphisms in the 8q24 locus. In addition, a genome-wide association study has completed. Statistical analyses of the questionnaire data are continuing.

ELIGIBILITY:
* INCLUSION CRITERIA:

The identification of men who have had a diagnosis of testicular germ cell tumor (TCGT) will be accomplished by the linking of databases maintained by the Department of Defense. Potential cases will be initially identified through the Defense Medical Surveillance System (DMSS).

Matched controls will be identified through the DMSS.

Criteria for Cases include:

Age between 17 and 45 years at time of confirmed TGCT diagnosis.

Age of at least 18 years at time of study enrollment.

The existence of a pre-diagnostic serum sample of 1mL or greater in the DoDSR.

On active duty at time of diagnosis.

Donated a serum sample to the DoDSR between the years 1989 and 2003.

Criteria for Control Identification:

Case subjects will be matched with case men on age, ethnicity, and date of serum donation to men in the DoDSR who have never had a diagnosis of TGCT (control men).

Criteria for Control Men include:

No previous diagnosis of TGCT.

Donated a serum sample to the DpDSR between the years 1989 and 2003.

Alive at study initiation.

On active duty at time of case's diagnosis.

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male U.S. servicemen, age 18-45 years old, with atleast one serum sample stored in the DoD Serum Repository.
Sampling Method: Non-Probability Sample
Enrollment: 2772 (Actual)
Dates: Start 2002-01-18 (Actual); Primary Completion 2008-10-01 (Actual); Study Completion 2020-08-18 (Actual)

PRIMARY OUTCOMES:
environmental and genetic determinants of TGCT risk | 16 years

CONTACTS AND LOCATIONS:
Overall Officials: Katherine A McGlynn, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Cancer Institute (NCI), 9000 Rockville Pike, Bethesda, Maryland, United States